CLINICAL TRIAL: NCT00500370
Title: A Pilot Study of Effects of Exenatide on Body Weight in Non-Diabetic, Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H8O-MC-GWBP
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
Keywords: exenatide; obesity; diabetes; Amylin; Lilly
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: exenatide
- Group B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide — subcutaneous injection (5mcg or 10mcg), twice a day
  Other Names: Byetta
  Arms: Group A
Drug: placebo — subcutaneous injection (equivalent volume to active dose), twice a day
  Arms: Group B

SUMMARY:
This is a multicenter study designed to compare the effect of exenatide plus a lifestyle modification plan versus placebo plus a lifestyle modification plan on weight loss in non-diabetic, obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index (BMI) >= 30kg/m^2

Exclusion Criteria:

* Have ever participated in this study previously, or any other study using exenatide (AC2993/LY2148568) or GLP-1 analogs
* Have participated in an interventional medical, surgical, or pharmaceutical study (a study in which an experimental, drug, medical, or surgical treatment was given) within 30 days of study start (this criterion includes drugs that have not received regulatory approval for any indication at the time of study entry)
* Diagnosis of diabetes mellitus (other than gestational diabetes), or previous use of anti-diabetic medications for > 3 months
* Have had a change in prescribed lipid-lowering or blood pressure agents within 4 weeks of screening
* Used drugs for weight loss (e.g., Xenical [orlistat], Meridia [sibutramine], Acutrim [phenylpropanolamine], Accomplia [rimonabant], Alli [low-dose orlistat], or other similar over-the-counter weight loss remedies or medications) within 3 months of screening
* Are actively participating in, or have participated in a formal weight loss program within the last 3 months
* Have a history of chronic use of drugs that directly affect gastrointestinal motility, including, but not limited to Reglan (metoclopramide) and chronic macrolide antibiotics
* Have been treated with any anti-diabetic medications within 3 months of screening
* Are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy or have received such therapy within the 4 weeks immediately prior to study start
* Have had bariatric surgery
* Have had an organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (16):
- United States (14):
  - Research Site, Peoria, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Santa Ana, California
  - Research Site, Indianapolis, Indiana
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, St Louis, Missouri
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Goose Creek, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Renton, Washington
- Puerto Rico (2):
  - Research Site, Ponce
  - Research Site, San Juan

REFERENCES:
- [Derived] Rosenstock J, Klaff LJ, Schwartz S, Northrup J, Holcombe JH, Wilhelm K, Trautmann M. Effects of exenatide and lifestyle modification on body weight and glucose tolerance in obese subjects with and without pre-diabetes. Diabetes Care. 2010 Jun;33(6):1173-5. doi: 10.2337/dc09-1203. Epub 2010 Mar 23. PMID 20332357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred between July 2007 and August 2007 at medical clinics in the United States.
Pre-assignment Details: Prior to randomization, subjects participated in a 1-week, single-blind placebo lead-in period.
Groups:
- Group A (Exenatide): exenatide 5mcg twice daily for 4 weeks plus lifestyle modification plan (LMP), followed by exenatide 10mcg twice daily for 20 weeks plus LMP
- Group B (Placebo): placebo (volume equivalent to exenatide injection) twice daily for 24 weeks plus LMP
Period: Overall Study
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Started | 80 | 83
Treatment Start-Baseline (Week 0) | 73 | 79
Treatment Complete (Week 24) | 48 | 54
Completed | 47 (COMPLETED = completion of treatment period (Week 24) plus follow-up visit 4 weeks later) | 49 (COMPLETED = completion of treatment period (Week 24) plus follow-up visit 4 weeks later)
Not Completed | 33 | 34
Not completed — Adverse Event | 9 | 3
Not completed — Lost to Follow-up | 10 | 10
Not completed — Protocol Violation | 2 | 4
Not completed — Sponsor Decision | 2 | 0
Not completed — Subject Decision | 10 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Exenatide) | Group B (Placebo) | Total
Number analyzed (Participants) | 73 | 79 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.01 (10.95) | 45.15 (12.74) | 46.04 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 67 | 125
  Male | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Change in body weight from baseline after 24 weeks of treatment (i.e., body weight at week 24 minus body weight at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 73 | 78
kg
  Baseline (Week 0) | 109.48 (2.70) | 107.64 (2.61)
  Change at Endpoint (Week 24) | -5.06 (0.49) | -1.61 (0.47)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures ANCOVA

2. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in BMI from baseline after 24 weeks of treatment (i.e., BMI at week 24 minus BMI at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 73 | 78
kg/m^2
  Baseline (Week 0) | 39.64 (0.82) | 39.39 (0.79)
  Change at Endpoint (Week 24) | -1.83 (0.18) | -0.58 (0.17)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures ANCOVA

3. Secondary Outcome: Change in Waist-to-hip Ratio
Description: Waist-to-hip ratio at week 24 compared to waist-to-hip ratio at week 0 (i.e., waist-to-hip ratio at week 24 minus waist-to-hip ratio at week 0). Waist-to-hip ratio equals waist circumference at given time point divided by hip circumference at given timepoint.
Time Frame: 24 weeks
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 69 | 70
Ratio
  Baseline (Week 0) | 0.90 (0.01) | 0.90 (0.01)
  Change at Endpoint (Week 24) | -0.001 (0.01) | 0.002 (0.01)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p = 0.6766, Mixed Model Repeated Measures ANCOVA

4. Secondary Outcome: Percentage of Patients Experiencing >=5% Weight Loss
Description: Percentage of exenatide and placebo treated patients experiencing >=5% weight loss after 24 weeks of treatment (i.e., [weight at week 0 minus weight at week 24] divided by weight at week 0 times 100% >=5%)
Time Frame: 24 weeks
Population: Intent to Treat population; Last Observation Carried Forward
Measure: Number; unit: percentage of patients
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 73 | 79
percentage of patients | 31.5 | 16.5
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.0393, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol from baseline after 24 weeks of treatment (i.e., total cholesterol at week 24 minus total cholesterol at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 67 | 70
mmol/L
  Baseline (Week 0) | 4.87 (0.11) | 4.88 (0.10)
  Change at Endpoint (Week 24) | 0.19 (0.11) | 0.33 (0.11)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p = 0.1808, ANCOVA

6. Secondary Outcome: Change in High Density Lipoprotein (HDL) Cholesterol
Description: Change in HDL cholesterol from baseline after 24 weeks of treatment (i.e., HDL cholesterol at week 24 minus HDL cholesterol at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 67 | 70
mmol/L
  Baseline (Week 0) | 1.27 (0.04) | 1.36 (0.04)
  Change at Endpoint (Week 24) | 0.004 (0.03) | 0.06 (0.03)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p = 0.1204, ANCOVA

7. Secondary Outcome: Ratio of Endpoint (LOCF) to Baseline for Fasting Triglycerides (Logarithmically Transformed)
Description: Ratio of triglycerides at week 24 compared to triglycerides at week 0 (i.e., triglycerides at week 24 divided by triglycerides at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 67 | 70
Ratio | 0.99 (0.06) | 0.96 (0.06)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.6651, ANCOVA

8. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol
Description: Change in LDL cholesterol from baseline following 24 weeks of treatment (i.e., LDL cholesterol at week 24 minus LDL cholesterol at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 67 | 67
mmol/L
  Baseline (Week 0) | 2.86 (0.10) | 2.79 (0.10)
  Change at Endpoint (Week 24) | 0.20 (0.09) | 0.34 (0.09)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p = 0.1204, ANCOVA

9. Secondary Outcome: Change in Fasting Serum Glucose
Description: Change in fasting serum glucose from baseline following 24 weeks of treatment (i.e., fasting serum glucose at week 24 minus fasting serum glucose at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 67 | 64
mmol/L
  Baseline (Week 0) | 5.37 (0.07) | 5.37 (0.07)
  Change at Endpoint (Week 24) | 0.000 (0.10) | -0.02 (0.10)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p = 0.8479, Mixed Model Repeated Measures ANCOVA

10. Secondary Outcome: Change in Serum Glucose AUC Levels Following Oral Glucose Tolerance Test (OGTT)
Description: Change in serum glucose AUC following OGTT (week 24 compared to week 0) (i.e., serum glucose AUC at week 24 minus serum glucose AUC at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: (mmol*hr)/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 62 | 62
(mmol*hr)/L
  Baseline (Week 0) | 15.73 (0.42) | 15.19 (0.42)
  Change at Endpoint (Week 24) | -0.47 (0.37) | -0.01 (0.37)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p = 0.2151, ANCOVA

11. Secondary Outcome: Ratio of Endpoint (LOCF) to Baseline for Homeostatic Model Assessment-Beta Cell (HOMA-B) (Logarithmically Transformed)
Description: Ratio of HOMA-B at week 24 to HOMA-B at week 0 (i.e., HOMA-B at week 24 divided by HOMA-B at week 0). HOMA-B is a measure of beta cell function.
Time Frame: 24 weeks
Population: Intent to Treat population; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 57 | 54
Ratio | 1.06 (0.07) | 1.08 (0.07)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.7619, ANCOVA

12. Secondary Outcome: Ratio of Endpoint (LOCF) to Baseline for Homeostatic Model Assessment-Insulin Sensitivity (HOMA-S) (Logarithmically Transformed)
Description: Ratio of HOMA-S at week 24 to HOMA-S at week 0 (i.e., HOMA-S at week 24 divided by HOMA-S at week 0). HOMA-S is a measure of insulin sensitivity.
Time Frame: 24 weeks
Population: Intent to Treat population; Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 57 | 54
Ratio | 0.92 (0.08) | 0.91 (0.08)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.8973, ANCOVA

13. Secondary Outcome: Incidence of Patients That Demonstrate Overt Signs of Diabetes Mellitus Diagnosis
Description: Number of patients in each treatment group that demonstrate overt signs of diabetes mellitus diagnosis by week 24
Time Frame: 24 weeks
Population: Intent to Treat population
Measure: Number; unit: Participants
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 65 | 65
Participants | 3 | 2
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.6507, Cochran-Mantel-Haenszel

14. Secondary Outcome: Incidence of Patients That Demonstrate Normalization of Impaired Fasting Glucose (IFG) and/or Impaired Glucose Tolerance (IGT)
Description: Number of patients in each treatment group that demonstrate normalization of IFG and/or IGT by week 24
Time Frame: 24 weeks
Population: Intent to Treat population
Measure: Number; unit: Participants
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 17 | 16
Participants | 13 | 9
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.2593, Cochran-Mantel-Haenszel

15. Secondary Outcome: Change in High Sensitivity C-reactive Protein (hsCRP)
Description: Change in hsCRP levels from baseline following 24 weeks of treatment (i.e., hsCRP at week 24 minus hsCRP at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 68 | 70
pmol/L
  Baseline (Week 0) | 8.61 (0.91) | 8.03 (0.90)
  Change at Endpoint (Week 24) | -1.31 (0.85) | -0.44 (0.83)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p = 0.2919, Mixed Model Repeated Measures ANCOVA

16. Secondary Outcome: Change in Glycosylated Hemoglobin (HbA1c)
Description: Change in HbA1c from baseline following 24 weeks of treatment (i.e., HbA1c at week 24 minus HbA1c at week 0)
Time Frame: 24 weeks
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 67 | 70
percent
  Baseline (Week 0) | 5.61 (0.04) | 5.58 (0.04)
  Change at Endpoint (Week 24) | -0.003 (0.04) | 0.09 (0.04)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Analysis pertains to change at endpoint (Week 24); Test type: Superiority or Other; p = 0.0293, Mixed Model Repeated Measures ANCOVA

ADVERSE EVENTS:
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/79
Other Adverse Events (participants affected / at risk) | 60/73 | 53/79
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Exenatide) (N=73) | Group B (Placebo) (N=79)
Nausea (Gastrointestinal disorders) | 18 | 3
Diarrhea (Gastrointestinal disorders) | 10 | 2
Headache (Nervous system disorders) | 7 | 5
Sinusitis (Infections and infestations) | 7 | 7
Vomiting (Gastrointestinal disorders) | 6 | 1
Pain (General disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dizziness (Nervous system disorders) | 4 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 0
Nasopharyngitis (Infections and infestations) | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Injection site bruising (General disorders) | 1 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days